CLINICAL TRIAL: NCT07262866
Title: Effect of Education and Counseling Provided Via Telenursing on Medication Compliance and Patient Satisfaction After Cataract Surgery
Brief Title: Evaluation of the Effects of Education and Counseling Provided to Patients Via Distance Nursing After Cataract Surgery on Regular Use of Medications and Patient Satisfaction. CAT-TELEMED (Cataract - Telemedicine) TNCat-25 (Tele-Nursing Cataract - 2025)
Acronym: TELE-NURSİNG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Züleyha Sönmez (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Züleyha Sönmez, research assistant, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/587
Record Dates: First submitted 2025-11-21; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Cataract Patients; Cataract After Surgery; Cataract Surgery
Keywords: Cataract; Cataract surgery; tele-nursing
MeSH Terms: conditions — Cataract | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: This study uses a parallel design in which participants are randomly assigned to one of two groups: an intervention group receiving structured tele-nursing education and counseling, and a control group receiving standard postoperative care. The groups are followed simultaneously throughout the study period without crossover.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-nursing Education (Experimental): Patients receive structured tele-nursing education and counseling through scheduled phone calls on postoperative days 1, 7, 15, and 30. The education includes medication adherence, eye care, symptom and complication management, nutrition, and balance precautions. Daily SMS(Short Message Service) reminders are sent during the first postoperative week to support medication adherence, followed by twice-weekly SMS (Short Message Service) reminders during weeks 2 to 4.
  Interventions: Behavioral: Structured Tele-Nursing Education and Counseling
- Standard Postoperative Care (No Intervention): Patients receive standard postoperative care without tele-nursing education or SMS (Short Message Service) reminders. They are contacted by phone once weekly for general follow-up during the first postoperative month.

INTERVENTIONS:
Behavioral: Structured Tele-Nursing Education and Counseling — This intervention is distinguished by its use of a combined tele-nursing approach involving scheduled telephone counseling and frequent SMS (Short Message Service) reminders to enhance medication adherence and patient satisfaction after cataract surgery. It provides continuous, personalized remote support focusing on symptom management, complication awareness, nutrition, and medication compliance over a 30-day postoperative period. Unlike traditional care models that rely on in-person visits or infrequent follow-ups, this intervention integrates real-time communication with automated reminders, improving patient engagement and outcomes.
  Other Names: Tele-Nursing Follow-up Program; Postoperative Remote Counseling; Cataract Surgery Tele-Care
  Arms: Tele-nursing Education

SUMMARY:
This randomized controlled study aims to investigate the effects of tele-nursing-based education and counseling on medication adherence and patient satisfaction following cataract surgery.

Cataract surgery is a common procedure, especially among the elderly, to improve visual function. However, the postoperative period is critical, and the success of the treatment greatly depends on whether patients use their prescribed eye drops and medications correctly and consistently. Patient satisfaction with the healthcare experience also plays a key role in overall outcomes.

The main hypothesis of this study is that structured education and counseling provided remotely by nurses (tele-nursing) will lead to better medication adherence and higher satisfaction compared to standard postoperative care.

Participants undergoing cataract surgery will be randomly assigned into two groups:

Intervention group: Will receive tele-nursing education and counseling via scheduled phone calls.

Control group: Will receive routine postoperative care with no additional support.

Nurses in the intervention group will educate patients on medication usage, eye care, possible complications, and other relevant topics after surgery. Follow-up calls will allow patients to ask questions and receive continuous support.

Both medication adherence and patient satisfaction will be measured using validated scales. Data will be analyzed using SPSS (Statistical Package for the Social Sciences) statistical software.

The results of this study may demonstrate the potential benefits of integrating tele-health interventions into postoperative care, especially in ophthalmology. It may also highlight the critical role of nurses in delivering remote patient education and support, contributing to the growing field of digital health.

DETAILED DESCRIPTION:
This randomized controlled study investigates the impact of tele-nursing education and counseling on medication adherence and patient satisfaction following cataract surgery.

Cataract surgery is a widely performed procedure to restore vision by replacing the eye's clouded lens. While the surgical technique is well established, postoperative management remains critical for successful outcomes. Patients must adhere to prescribed eye drops and medications to prevent infection, control inflammation, and promote healing. Non-adherence can increase the risk of complications such as infection or poor visual recovery.

The study tests the hypothesis that structured, nurse-led telephonic education and counseling improves medication adherence and enhances patient satisfaction compared to standard postoperative care.

Participants who have undergone cataract surgery are randomly allocated to either:

An intervention group receiving scheduled tele-nursing sessions that provide education on medication administration, eye care, signs of complications, and emotional support.

A control group receiving routine postoperative instructions without additional tele-nursing support.

Tele-nursing sessions are designed to be interactive, allowing patients to ask questions and receive tailored advice. This method leverages accessible technology (telephone) to overcome barriers like geographical distance, mobility limitations, or lack of in-person follow-up resources.

Data collection focuses on self-reported medication adherence and validated patient satisfaction questionnaires, analyzed statistically to determine the effectiveness of tele-nursing interventions.

This study contributes evidence on integrating telehealth approaches in postoperative care protocols, potentially offering scalable solutions to improve patient outcomes and healthcare quality in ophthalmology.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients who voluntarily agree to participate in the study
* Patients able to communicate in Turkish
* Patients who own a personal mobile phone
* Patients who can read text messages or have a relative at home who can assist them after discharge
* Patients without hearing impairments
* Patients undergoing eye surgery (cataract surgery) for the first time

Exclusion Criteria:

* Patients under 18 years of age
* Patients who do not volunteer to participate in the study
* Patients who do not understand Turkish and cannot communicate in Turkish
* Patients with any psychiatric illness
* Patients with hearing or perception problems

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale - Satisfaction (VAS-S) | Postoperative day 30
  Patient satisfaction will be assessed using the Visual Analog Scale - Satisfaction (VAS-S). This scale ranges from 0 to 10, where: 0 = No satisfaction, 10 = Highest possible satisfaction. Higher scores indicate better patient satisfaction
Medication Adherence Reporting Scale | Postoperative day 30
  Medication adherence will be evaluated using the Medication Adherence Self-Report Scale, a 5-item, 5-point Likert-type self-report scale.
  The scale total score ranges from 5 to 25, where: 5 = Lowest medication adherence, 25 = Highest medication adherence, Higher scores indicate better medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞEGÜL YAYLA, ASSOCIATE PROFESSOR, Principal Investigator — Ataturk University; WORK Ataturk University, Principal Investigator — Atatürk Üniversitesi 25240 Erzurum/ TURKEY
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) from this randomized controlled trial will be shared with qualified researchers for academic or clinical research purposes. Shared data will include de-identified demographic information, treatment allocation, and outcome measurements. Data will be available after publication of the primary results. Access will be granted upon request through a data-sharing agreement to ensure confidentiality and ethical use.